CLINICAL TRIAL: NCT02405364
Title: Front-line Therapy With Carfilzomib, Lenalidomide, and Dexamethasone (CRd) Induction Followed by Autologous Stem Cell Transplantation, CRd Consolidation and Lenalidomide Maintenance in Newly Diagnosed Multiple Myeloma Patients ≤65 Years Old
Brief Title: Front-line Therapy With Carfilzomib, Lenalidomide, and Dexamethasone Induction
Acronym: IFM-CRd
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Onyx Therapeutics, Inc. (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12 568 03
Record Dates: First submitted 2013-10-16; First posted 2015-04-01 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Carfilzomib; Lenalidomide; Dexamethasone; Patient up to 65 years; initial management
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- Front line therapy (Experimental): Induction: 4 cycles of 28 days of Carfilzomib/Lenalidomide/Dexamethasone Stem Cell Harvest+Intensification Consolidation 4 cycles of 28 days of Carfilzomib/ Lenalidomide/Dexamethasone Maintenance: Lenalidomide 13 cycles of 28 days
  Interventions: Drug: Carfilzomib/Lenalidomide/Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib/Lenalidomide/Dexamethasone — Induction:Carfilzomib/Lenalidomide/Dexamethasone (4 cycles every 28 days) Stem Cell harvest: HD Cyclophosphamide Intensification: HD Melphalan Consolidation:Carfilzomib/Lenalidomide/Dexamethasone (4 cycles every 28 days) Maintenance: Lenalidomide (13 cycles)
  Other Names: New drug combination

SUMMARY:
The purpose is to determine whether induction and consolidation treatment with Carfilzomib, Lenalidomide and Dexamethasone (CRd), within an intensive program, warrant further investigation in clinical trials.

DETAILED DESCRIPTION:
The primary objective is to evaluate the sCR rate of the combination of carfilzomib, lenalidomide and dexamethasone in newly diagnosed multiple myeloma patients at the completion of consolidation therapy.

It's a multicenter, open label, non randomized, phase II study. 46 patients will be enrolled.

Induction: 4 cycles of 28 Days with Carfilzomib/Lenalidomide and dexamethasone Stem Cell Harvest: High dose Cyclophosphamide with intensification consolidation: 4 cycles of 28 Days with Carfilzomib/Lenalidomide and dexamethasone Maintenance : Lenalidomide 13 cycles of 28 days

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with multiple myeloma based on the new International Myeloma Working Group
* Subjects must have symptomatic myeloma with at least one CRAB criteria
* Subjects must not have been treated previously with any systemic therapy for multiple myeloma

Exclusion Criteria:

* Pregnant or lactating females
* Evidence of mucosal or internal bleeding and/or platelet refractory
* Acute active infection requiring treatment
* Treatment by localized radiotherapy if the interval between the end of radiotherapy and initiation of protocol therapy lower than 2 weeks
* Treatment by corticosteroids if exceed the equivalent of 160 mg of dexamethasone in a 2-week period before initiation therapy
* Subjects not eligible for high dose therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
rate of stringent complete response | 12 months
  completion of consolidation

CONTACTS AND LOCATIONS:
Overall Officials: Michel ATTAL, MD, Principal Investigator — University Hospital of Toulouse; Murielle ROUSSEL, MD, Principal Investigator — University Hospital of Toulouse
Locations (11):
- France (11):
  - CHU Henri Mondor, Créteil
  - CHRU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - Hôpital Claude Huriez, Lille
  - CHRU Hôtel Dieu, Nantes
  - Hôpital Saint-Antoine, Paris
  - Hôpital de Pontchaillou, Rennes
  - Hôpital de Hautepierre, Strasbourg
  - CHU de Toulouse, Toulouse
  - University hospital of Toulouse, Toulouse
  - Hôpital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Landgren O, Kazandjian D, Roussel M, Jasielec J, Dytfeld D, Anderson A, Kervin TA, Iskander K, McFadden I, Jakubowiak AJ. Efficacy and safety of carfilzomib-lenalidomide-dexamethasone in newly diagnosed multiple myeloma: pooled analysis of four single-arm studies. Leuk Lymphoma. 2022 Oct;63(10):2413-2421. doi: 10.1080/10428194.2022.2068001. Epub 2022 May 12. PMID 35549810
- [Derived] Roussel M, Lauwers-Cances V, Wuilleme S, Belhadj K, Manier S, Garderet L, Escoffre-Barbe M, Mariette C, Benboubker L, Caillot D, Sonntag C, Touzeau C, Dupuis J, Moreau P, Leleu X, Facon T, Hebraud B, Corre J, Attal M. Up-front carfilzomib, lenalidomide, and dexamethasone with transplant for patients with multiple myeloma: the IFM KRd final results. Blood. 2021 Jul 15;138(2):113-121. doi: 10.1182/blood.2021010744. PMID 33827114